CLINICAL TRIAL: NCT05240248
Title: Assessment of Optilene® Suture Material for Skin Closure (Dermal Sutures). A Prospective Single-arm Observational Study in Daily Practice
Brief Title: Optilene® Suture Material for Dermal Sutures
Acronym: OPTIDERMAL
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1928
Record Dates: First submitted 2022-01-26; First posted 2022-02-15 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Laceration; Incision
MeSH Terms: conditions — Lacerations; Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this non-interventional study, Optilene® suture will be evaluated for skin closure in adult patients.

DETAILED DESCRIPTION:
The study is designed as a prospective, unicentric and single-arm observational study to evaluate Optilene® suture material for skin closure.

The product under investigation will be used in routine clinical practice and according to the Instructions for Use (IFU). After operation the investigator will examine the patients at discharge, at 10±5 days after surgery (removal of the suture) and 30±10 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing skin closure using Optilene® suture material.
* Small (0.5 cm - 10 cm) linear minimally contaminated incision/laceration in the trunk, neck or extremities (in the event that more than one incision is performed in the same patient, only one incision will be included).
* Written informed consent.

Exclusion Criteria:

* Emergency surgery.
* Transplant surgery.
* Pregnancy.
* Facial laceration or incision.
* Visible dirt in the wound.
* Non-linear shape.
* Patient with limb ischemia.
* Patient taking medication that might affect wound healing (i.e. cytotoxic antineoplastic and immunosuppressive agents, corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), anticoagulants).
* Patient with hypersensitivity or allergy to the suture material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing skin closure using Optilene® suture material.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | at suture removal approximately 10±5 days postoperatively.
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections involving the skin only. Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material.

SECONDARY OUTCOMES:
Surgical Site Infection Rate | at discharge from hospital (up to 5 days postoperatively)
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections involving the skin only. Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material.
Surgical Site Infection Rate | at follow-up examination approximately 30±10 days postoperatively
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections involving the skin only. Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material.
Wound dehiscence rate | at discharge from hospital (up to 5 days postoperatively)
  Pathologic process consisting of a partial or complete disruption of the layers of a surgical wound.
Wound dehiscence rate | at suture removal approximately 10±5 days postoperatively.
  Pathologic process consisting of a partial or complete disruption of the layers of a surgical wound.
Wound dehiscence rate | at follow-up examination approximately 30±10 days postoperatively
  Pathologic process consisting of a partial or complete disruption of the layers of a surgical wound.
Cumulative rate of Adverse Events during the study period | at discharge (up to 5 days postoperatively), at suture removal (approximately 10±5 days postoperatively) and at follow-up visit approximately 30±10 days postoperatively
  frequency of Tissue reaction, Inflammation, Seroma, Abscess formation, Hematoma, Granuloma, Bleeding, Necrosis and Irritation
Development of Cosmetic Outcome | at discharge (up to 5 days postoperatively), at suture removal (approximately 10±5 days postoperatively) and at follow-up visit approximately 30±10 days postoperatively
  Overall patient and observer satisfaction with the scar using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome in six categories (Pain, Itching, Color of scar, Stiffness of scar, thickness and irregularity of scar) on a 1 to 10 points scale each. The physician will use the Observer component, rating vascularization, pigmentation, thickness, relief and pliability of the scar on a 1 to 10 points scale each. The categories are added to a total POSAS score of 11 (minimum) to 110 points (maximum).
Development of Pain: Visual Analogue Scale (VAS) | at suture removal (approximately 10±5 days postoperatively) and at follow-up visit approximately 30±10 days postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".
Development of Satisfaction of the patient: Visual Analogue Scale (VAS) | at suture removal (approximately 10±5 days postoperatively) and at follow-up visit approximately 30±10 days postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "very poor" and "100" at the opposite end representing "excellent".
Duration of surgery | intraoperatively
  time from cut to closure in minutes.
Handling of the suture material | intraoperatively
  The handling of the suture material is assessed using a questionnaire assessing the Knot security (The quality of a suture that allows it to be tied securely with a minimum number of throws per knot), the Knot pull tensile strength (strength of the thread while knotting), the Knot run down (Ease with which a knot can be slid down), the Tissue drag (Passage through the tissue), the Pliability (The quality of being easily to bent, flexibility) and the Overall opinion of the surgeon each with the 5 evaluation levels of 'excellent', 'very good', 'good', 'satisfied' and 'poor':.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Doctor Peset, Valencia, Spain